CLINICAL TRIAL: NCT00114959
Title: A Phase II Open-Label Study of the Intravenous Administration of Homoharringtonine (CGX-635) Combined With the Oral Administration of Gleevec in the Treatment of Patients With Chronic Myeloid Leukemia (CML) in Chronic, Accelerated, and Blast Phase
Brief Title: Homoharringtonine With Oral Gleevec in Chronic, Accelerated and Blast Phase Chronic Myeloid Leukemia (CML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: ChemGenex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGX-635-CML-201; MDACC protocol #2005-0067 (Other: M.D. Anderson Cancer Center)
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Myeloid Leukemia, Chronic; Myeloid Leukemia, Chronic, Accelerated-Phase; Blast Phase; Myeloid Leukemia, Chronic, Chronic-Phase
Keywords: ChemGenex Pharmaceuticals, Ltd; ChemGenex Pharmaceuticals; ChemGenex; Chronic Myeloid Leukemia; Myeloid Leukemia, Chronic; Leukemia; Myeloid Leukemia; Chronic Phase; Accelerated Phase; Blast Phase; Myeloid, Leukemia, Chronic, Accelerated Phase; Myeloid, Leukemia, Chronic; Leukemia, Myeloid, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Chronic Phase; Leukemia, Myeloid, Accelerated-Phase; Myeloid, Leukemia, Chronic, Chronic Phase; Leukemia, Myeloid, Accelerated Phase; Homoharringtonine; Omacetaxine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia; Leukemia, Myeloid | interventions — Homoharringtonine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Homoharringtonine + Imatinib Mesylate (Experimental): Participants are administered homoharringtonine (omacetaxine) 2.5 mg/m^2 by continuous 24-hour intravenous infusion daily on Days 1-5 of each 4 week treatment cycle, and imatinib mesylate (Gleevec) by mouth with a daily dose of 400 mg for participants in the chronic phase of chronic myeloid leukemia (CML) or 600 mg for participants in the accelerated or blast phase of CML.
  Interventions: Drug: Homoharringtonine; Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Homoharringtonine — Participants are administered homoharringtonine (omacetaxine) 2.5 mg/m^2 by continuous 24-hour intravenous (IV) infusion daily on Days 1-5 of each 4 week treatment cycle. Participants who do not achieve a meaningful hematologic or cytogenetic response by the end of the fourth cycle are discontinued from the study. Otherwise, participants may continue additional cycles of this combined treatment for a maximum of 12 cycles.
  Participants who achieved a molecular or cytogenetic response, or a complete hematologic remission (CHR), could undergo subsequent cycles with a maintenance schedule of homoharringtonine 2.5 mg/m^2 by continuous 24-hour IV infusion daily for 2 days every 4 weeks. Dose escalations in subsequent cycles were allowed by one day at a time if the participant was unable to maintain CHR in the maintenance schedule.
  Other Names: Omacetaxine mepesuccinate; CGX-635
Drug: Imatinib Mesylate — Taken by mouth with a daily dose of 400 mg for participants in the chronic phase of chronic myeloid leukemia (CML) or 600 mg for participants in the accelerated or blast phase of CML. For the first cycle of therapy only, imatinib was started on Day 4 of homoharringtonine treatment.
  Other Names: Gleevac

SUMMARY:
This will be an open label, multi-center study of up to 77 patients with CML in chronic, accelerated or blast phase who have developed resistance to or have failed previous treatment with Gleevec (imatinib mesylate). Because these patients may still be sensitive to Gleevec, adding Homoharringtonine may restore a response to Gleevec or the combined treatment may promote a better response than using Gleevec alone.

DETAILED DESCRIPTION:
Every 4 weeks, the study medicine Homoharringtonine will be given by vein daily for 5 days along with continuing daily doses of the approved medicine Gleevec taken by mouth. The safety and effectiveness of this combined treatment in CML patients will be studied. Patients who do not achieve a meaningful hematologic or cytogenetic response after 4 cycles or less will be discontinued. Otherwise, patients may continue additional cycles of this combined treatment for a maximum of 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 16 years or older
* Philadelphia chromosome (Ph) positive chronic myelogenous leukemia (CML) in either chronic, accelerated or blast phase
* Patients with chronic phase CML will be either refractory (failed to achieve hematologic or cytogenetic response) or resistant (responded initially but subsequently lost hematologic or cytogenetic response) to prior imatinib mesylate therapy. Failure to achieve cytogenetic response is defined as follows: no cytogenetic response after 3 months of therapy with imatinib mesylate, no major cytogenetic response at 12 months of therapy, loss of complete cytogenetic response documented twice, or loss of major cytogenetic response at least once.
* Patients with accelerated or blast phase may be newly diagnosed and previously untreated or if previously treated with imatinib mesylate, will be refractory or resistant to this agent or have failed to achieve at least a complete hematologic or cytogenetic response to treatment, as previously defined.
* Patients in accelerated phase will meet one or more of the following criteria: greater than or equal to 15% through less than 30% blasts in peripheral blood or bone marrow, greater than or equal to 30% blasts + promyelocytes in peripheral blood or bone marrow, greater than or equal to 20% basophils in peripheral blood, platelet count less than 100*10^9/L unrelated to therapy or clonal evolution.
* CML in blast phase will be defined as greater than or equal to 30% blasts in the bone marrow or presence of extramedullary disease
* Patients must have completed all previous anti-leukemic therapy for at least 2 weeks, except as noted, and have fully recovered from side effects of a previous therapy, unless disease progression necessitates early therapy. Patients may receive leukapheresis, hydroxyurea and anagrelide for up to 24 hours prior to start of study treatment. Patients receiving imatinib mesylate may continue to receive it uninterrupted, except for a 3-day window at treatment cycle 1.
* Bilirubin less than or equal to 2 times the upper limit of normal (ULN); alanine aminotransferase (ALT) less than or equal to 3 times ULN; creatinine less than or equal to 1.5 times ULN
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Be able to comply with the requirements of the entire study
* Be able and willing to provide written informed consent prior to any study related procedure
* Patients and their partners must use an effective contraceptive during the study dosing period. The following are considered effective contraceptives: oral contraceptive pill, condom, diaphragm plus spermicide, abstinence, patient or partner surgically sterile, patient or partner more than 2 years post-menopausal, or injectable or implantable agent/device.

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia and requiring therapy, uncontrolled hypertension or congestive heart failure
* Myocardial infarction in the previous 12 weeks
* Other intercurrent illness which would preclude study conduct and assessment, including but not limited to another active malignancy, uncontrolled and active infection, positive human immunodeficiency virus (HIV) or human T-cell lymphotropic virus (HTLV) I/II status
* Pregnant or lactating
* Any medical or psychiatric condition which may compromise the ability to give written informed consent or to comply with the study protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam R Craig, M.D., PhD, Study Director — ChemGenex Pharmaceuticals; Jorge Cortes, M.D., Principal Investigator — Univ. of TX M.D. Anderson Cancer Center
Locations (1):
- Univ. of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Homoharringtonine + Imatinib Mesylate
Started | 15
Completed | 7 (protocol definition of completed study is having received >= 4 cycles of treatment)
Not Completed | 8
Not completed — Lack of Efficacy | 6
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Homoharringtonine + Imatinib Mesylate
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 55 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 4
  Caucasian | 10
  Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Accelerated Phase or Blast Phase Chronic Myeloid Leukemia (CML) Who Achieve a Meaningful Response
Description: Participants in accelerated or blast phase who converted to at least CML-chronic phase.
  CML in accelerated phase meets one or more of the following criteria: >=15% - <30% blasts in peripheral blood or bone marrow, >=30% blasts + promyelocytes in peripheral blood or bone marrow, >=20% basophils in peripheral blood; platelet count <100*10^9/L unrelated to therapy or clonal evolution. CML in blast phase have >=30% blasts in the bone marrow or presence of extramedullary disease.
  Meaningful responses include (in descending order of health)
  * Complete Hematologic Remission (CHR)
  * Partial Hematologic Remission (PHR)
  * Hematologic Improvement (HI)
  * Partial Response (PR)
  * Return to Chronic Phase (RCP). A return to chronic phase involves the disappearance of blastic phase features and a return to chronic phase CML picture, i.e., peripheral blasts <15%, peripheral blasts and promyelocytes <30%, peripheral basophils <20%, and platelets >100*10^9/L.
Time Frame: up to month 4
Population: No participants were analyzed since the study was intended to follow a Simon two stage design to test 18 participants in each stratum (chronic, accelerated and blast phases) for efficacy. Enrollment was insufficient.
Arm/Group | Homoharringtonine + Imatinib Mesylate
Number analyzed (Participants) | 0

2. Primary Outcome: Proportion of Participants With Chronic Phase Chronic Myeloid Leukemia (CML) Who Achieve a Meaningful Response
Description: Participants who are not in complete hematologic remission (CHR) at study start must achieve at least a CHR, and participants who are in CHR at onset must demonstrate an improvement in their cytogenetics.
  A Complete Hematologic Remission (CHR) involves normalization of the bone marrow (less than 5% blasts) and peripheral blood with white blood cells < 10*10^9/L, absolute neutrophil count >=1*10^9/L, platelets >=100*10^9/L and no peripheral blasts, promyelocytes or myelocytes. This is in addition to disappearance of all signs and symptoms of the disease.
Time Frame: up to month 4
Population: as for outcome 1
Arm/Group | Homoharringtonine + Imatinib Mesylate
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Adverse Experiences (AEs)
Description: Summary of participants who had adverse events (AEs), who discontinued treatment due to the AE, who had serious adverse events (SAEs), and who had SAEs that were related to treatments.
  A serious adverse event is one that at any dose of the study drug or at any time during the period of observation:
  * Results in death;
  * Is life threatening;
  * Requires inpatient hospitalization or prolongation of existing hospitalization;
  * Results in persistent or significant disability/incapacity;
  * Is a congenital anomaly/birth defect;
  * Is medically important.
  The Investigator assessed each AE for potential causal relationship between the event and study drug. An investigator assessment of possibly, probably or unknown relation is considered related.
Time Frame: up to 3 years
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Homoharringtonine + Imatinib Mesylate
Number analyzed (Participants) | 15
participants
  AEs | 15
  Discontinued due to AE | 2
  Serious AEs | 12
  SAEs considered related | 7

4. Secondary Outcome: Participants With Complete Hematologic Remission Suppression of the Philadelphia Chromosome
Description: Complete hematologic remission was further classified according to the suppression of the Philadelphia chromosome (Ph) as:
  No cytogenetic response - Ph positive 100% Minimal cytogenetic response - Ph positive 35-90% Partial cytogenetic response - Ph positive 1-34% Complete cytogenetic response - Ph positive 0%
Time Frame: up to month 4
Population: as for outcome 1
Arm/Group | Homoharringtonine + Imatinib Mesylate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 3 years (30 days past last dose)
Arm/Group | Homoharringtonine + Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 12/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Homoharringtonine + Imatinib Mesylate (N=15)
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 3
Renal failure (Renal and urinary disorders) | 1
Pain, upper extremities (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 2
Infection (General disorders) | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 1
Hemorrhage, gastrointestinal (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fatal car accident (Injury, poisoning and procedural complications) | 1
Weakness (General disorders) | 1
Cerebral vascular event (fatal) (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Acute renal failure (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Intra-cranial hemorrhage (Vascular disorders) | 1
Sudden death (General disorders) | 1
Leukocytosis (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Death (General disorders) | 1
Pain, low back (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Homoharringtonine + Imatinib Mesylate (N=15)
Allergies (General disorders) | 1
Bacteremia (General disorders) | 1
Bleeding at CVC site (General disorders) | 1
Bleeding at PICC line insertion site (General disorders) | 1
Bleeding at port site (General disorders) | 1
Bruising (General disorders) | 2
Chills (General disorders) | 2
Chills, intermittent (General disorders) | 1
Citrobacter freundii positive (General disorders) | 1
Fatigue (General disorders) | 7
Mild fatigue (General disorders) | 4
Severe fatigue (General disorders) | 1
Fever (General disorders) | 2
Fibromyalgia syndrome (General disorders) | 1
Fluid retention (Gastrointestinal disorders) | 2
Generalized achiness (General disorders) | 1
Infection, Staphylococcus aureus (Infections and infestations) | 1
Intermittent fatigue (General disorders) | 1
Intermittent fever (General disorders) | 1
Mild fever (General disorders) | 1
Pain, left flank (General disorders) | 1
Pain, left upper quadrant (General disorders) | 1
Pain, right hip (General disorders) | 1
Pallor (General disorders) | 1
Pseudomonas aeruginosa (Infections and infestations) | 1
Runny nose (General disorders) | 1
Weakness (General disorders) | 1
Mildly weak (General disorders) | 1
Edema (General disorders) | 2
Edema, intermittent (General disorders) | 1
Edema, pedal (General disorders) | 1
Edema, ankle (General disorders) | 2
Edema, bilateral (General disorders) | 1
Edema, bilateral pedal (General disorders) | 1
Edema, bilateral legs + 2 pitting (General disorders) | 1
Edema, bilateral lower extremity (General disorders) | 3
Edema, lower extremity (General disorders) | 2
Edema, peripheral (General disorders) | 2
Edema, Intermittent trace peripheral (General disorders) | 1
Hemoglobin decreased (Investigations) | 1
Leukocytosis (Investigations) | 1
Palpitations (General disorders) | 1
Periorbital edema (General disorders) | 1
Right Arm Swelling (General disorders) | 1
Right side face swelling (General disorders) | 1
Severe thrombocytopenia (Investigations) | 1
Swelling, hands and feet (General disorders) | 1
Swelling, right arm (General disorders) | 1
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1
Bruising skin (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema, left foot (Skin and subcutaneous tissue disorders) | 1
Erythema, tonsils (Skin and subcutaneous tissue disorders) | 1
Hypopigmentation facial (Skin and subcutaneous tissue disorders) | 1
Itching due to transfusion (Skin and subcutaneous tissue disorders) | 1
Itching impaired (Skin and subcutaneous tissue disorders) | 1
Generalized skin itching (Skin and subcutaneous tissue disorders) | 2
Itchy ears (Skin and subcutaneous tissue disorders) | 1
Keratoderma, pedal (Skin and subcutaneous tissue disorders) | 1
Pedal calluses (Skin and subcutaneous tissue disorders) | 1
Mild rash (Skin and subcutaneous tissue disorders) | 1
Mouth sores (Skin and subcutaneous tissue disorders) | 1
Mouth sores, intermittent (Skin and subcutaneous tissue disorders) | 1
Mouth ulcerations (Skin and subcutaneous tissue disorders) | 1
Oral white patches (Skin and subcutaneous tissue disorders) | 1
Peeling skin, groin (Skin and subcutaneous tissue disorders) | 1
Plantar surface skin sensitive (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Painful, red, swollen rash (Skin and subcutaneous tissue disorders) | 1
Rash abdomen (Skin and subcutaneous tissue disorders) | 1
Rash, macular / facial (Skin and subcutaneous tissue disorders) | 1
Seborrheic keratosis, upper extremity (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Swelling, face (Skin and subcutaneous tissue disorders) | 1
Tinea (Skin and subcutaneous tissue disorders) | 1
Punctate lesion right foot dorsom (Skin and subcutaneous tissue disorders) | 1
Vesicular lesions, right buttock (Skin and subcutaneous tissue disorders) | 1
Yeast infection, buttock (Skin and subcutaneous tissue disorders) | 1
Abdominal bloating (Gastrointestinal disorders) | 1
Abdominal discomfort intermittent (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain, interrmittent left sided (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Colon polyps (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Constipation, intermittent (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dry heaves (Gastrointestinal disorders) | 1
Flatus (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
GERD (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hepatic Dysfunction (Gastrointestinal disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Lack of appetite (Gastrointestinal disorders) | 1
Poor appetite (Gastrointestinal disorders) | 2
Suppressed appetite (Gastrointestinal disorders) | 1
Loose stools (Gastrointestinal disorders) | 3
Melena (Gastrointestinal disorders) | 1
Mild nausea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Nausea, intermittent (Gastrointestinal disorders) | 1
Pandiverticulosis (Gastrointestinal disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Renal failure (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Upset stomach (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 11
Vomiting, occasional (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 9
Bruising (Blood and lymphatic system disorders) | 1
Abdominal bruising, secondary to SC injections (Blood and lymphatic system disorders) | 2
Decreased prothrombinemia (Blood and lymphatic system disorders) | 1
Ecchymoses, mouth and arms (Blood and lymphatic system disorders) | 1
Elevated BUN (Investigations) | 1
Elevated PTT (Investigations) | 1
Decreased hemaglobin (Investigations) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Hepatitis A (Blood and lymphatic system disorders) | 1
Hypertriglyceridemia (Blood and lymphatic system disorders) | 1
Intermittent anemia (Blood and lymphatic system disorders) | 1
Myelosuppression (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 8
Neutropenic fever (Blood and lymphatic system disorders) | 2
Nosebleed (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 3
Petechiae (Blood and lymphatic system disorders) | 2
Petechiae abdomen (Blood and lymphatic system disorders) | 1
Petechiae head, arms, neck, oral (Blood and lymphatic system disorders) | 1
Petechiae thigh (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia, intermittent (Blood and lymphatic system disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Elevated creatinine (Investigations) | 1
Elevated LDH (Investigations) | 1
Goiter, nodular (Metabolism and nutrition disorders) | 1
Hot flashes (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hypomagnesium (Metabolism and nutrition disorders) | 2
Uricemia (Metabolism and nutrition disorders) | 1
Aching all over (Musculoskeletal and connective tissue disorders) | 1
Bilateral upper pain - extremities (Musculoskeletal and connective tissue disorders) | 1
Cellulitis, left arm (Musculoskeletal and connective tissue disorders) | 1
Chest pain (Musculoskeletal and connective tissue disorders) | 1
Chest pressure (Musculoskeletal and connective tissue disorders) | 1
Cramps right leg, right arm (Musculoskeletal and connective tissue disorders) | 1
Cramps, muscle (Musculoskeletal and connective tissue disorders) | 1
Cramps, neck (Musculoskeletal and connective tissue disorders) | 1
Cramps, pedal muscle bilateral (Musculoskeletal and connective tissue disorders) | 1
Dental abscesses (Musculoskeletal and connective tissue disorders) | 1
Diffused bone pain (Musculoskeletal and connective tissue disorders) | 1
Left hip and leg pain, secondary to bone marrow aspiration (Musculoskeletal and connective tissue disorders) | 1
Leg muscle soreness (Musculoskeletal and connective tissue disorders) | 1
Leg trembling on standing (Musculoskeletal and connective tissue disorders) | 1
Pain, bilateral knee (Musculoskeletal and connective tissue disorders) | 1
Pain, bilateral shoulder (Musculoskeletal and connective tissue disorders) | 2
Pain, bone (Musculoskeletal and connective tissue disorders) | 2
Pain, knee (Musculoskeletal and connective tissue disorders) | 1
Pain, left knee (Musculoskeletal and connective tissue disorders) | 1
Pain, left great toe (Musculoskeletal and connective tissue disorders) | 1
Pain, low back (Musculoskeletal and connective tissue disorders) | 1
Pain, muscle (Musculoskeletal and connective tissue disorders) | 1
Pain, back and shoulder (Musculoskeletal and connective tissue disorders) | 1
Pain, neck (Musculoskeletal and connective tissue disorders) | 1
Pain, upper extremities (Musculoskeletal and connective tissue disorders) | 1
Teeth sensitivity (Musculoskeletal and connective tissue disorders) | 1
Tooth pain (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Nervous system disorders) | 1
Bad dreams (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Mild confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dizziness, fentanyl (Nervous system disorders) | 1
Dysphagia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Headache/migraine, intermittent right side (Nervous system disorders) | 1
Headache, sinus (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 1
Light headed (Nervous system disorders) | 2
Neuropathy, bipedal (Nervous system disorders) | 1
Neuropathy, hands and feet (Nervous system disorders) | 1
Peripheral neuropathy, secondary to diabetes (Nervous system disorders) | 1
Night sweats (Nervous system disorders) | 2
Numbness, toe (Nervous system disorders) | 1
Numbness/tingling in extremities (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Klebsiella pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
Short of breath (Respiratory, thoracic and mediastinal disorders) | 2
Shortness of breath on exertion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion intermittent, secondary to allergies (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory infection nasal allergies (Respiratory, thoracic and mediastinal disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Bleeding gums (General disorders) | 4
Conjunctival melanosis (Eye disorders) | 1
Dental extraction (Surgical and medical procedures) | 1
Gum soreness (General disorders) | 1
Gum tenderness (General disorders) | 1
Itchy eyes (Eye disorders) | 1
Lip bleeding (General disorders) | 1
Loss of taste (General disorders) | 1
Malodor, secondary to right groin hematoma (General disorders) | 1
Mucositis (General disorders) | 1
Oral ulcer (General disorders) | 1
Right Ear Pressure (General disorders) | 1
Sinus drainage (General disorders) | 1
Staph infection right nostril (Infections and infestations) | 1
Throat pain (General disorders) | 1
Worsening otitis media (Ear and labyrinth disorders) | 1
Dark urine (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 3

LIMITATIONS AND CAVEATS:
This study was intended to follow a Simon two stage design to test 18 patients in each stratum (chronic, accelerated and blast phase) for efficacy. Only 15 were enrolled, an insufficient number for a formal statistical analysis of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.